

| BI Study Number: 1199.402 | |
|---|---|
| Title: | Post-marketing Surveillance of Ofev Capsules in Chronic fibrosing Interstitial Lung Diseases with a progressive phenotype in Japan |
| NCT number: | NCT04559581 |
| Date: | 15-Mar-2025 |

This page has been added to the Statistical and Epidemiological Analysis Plan (SEAP) to reflect the requirements by ClinicalTrials.gov. This information is not part of the standard document.



### Global ID:228892\_82584\_1.0

| <del>_</del> | <del>-</del> |
|---|---|
| Document Number: | VV-TMF-82584 |
| BI Study Number: | 1199.402 |
| BI Investigational<br>Product(s) | Nintedanib |
| Title: | Post-marketing Surveillance of Ofev Capsules in Chronic fibrosing Interstitial Lung Diseases with a progressive phenotype in Japan |
| Brief lay title: | PMS of Ofev Capsules in PF-ILD |
| SEAP version identifier: | Version 1.0 |
| Date of last version of SEAP: | NA |
| ONIS Statistician [SEAP author] | |
| ONIS [SEAP reviewer] | |
| ONIS Data [SEAP reviewer] | |

Proprietary confidential information © 2025 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

### **TABLE OF CONTENTS**

| 1. L | LIST OF ABBREVIATIONS | 3 |
|-------------|----------------------------------------------------|---|
| 2. F | RESPONSIBLE PARTIES | 4 |
| | PURPOSE AND SCOPE | |
| 4. <i>A</i> | AMENDMENTS AND UPDATES | 4 |
| 5. F | RESEARCH QUESTION AND OBJECTIVE | 4 |
| 6. F | RESEARCH METHODs | 5 |
| 6.1 | STUDY DESIGN | 5 |
| 6.2 | | |
| 6.2 | J | |
| 6.2 | 2.2 Inclusion/ exclusion criteria | |
| 6.2 | 2.3 Registration period | |
| 6.2 | Patient registration method | 5 |
| 6.3 | STUDY POPULATION | |
| 6.4 | STUDY VISITS | |
| | VARIABLES | |
| 7.1 | EXPOSURES | |
| 7.2 | OUTCOMES | |
| | Primary outcomes | |
| 7.2 | 2.2 Secondary outcomes | 9 |
| 7.3 | | |
| | DATA SOURCES 1 | |
| | DATA MANAGEMENT and Software/Tools | |
| 9.1 | SOFTWARE/TOOLS | |
| 9.2 | HANDLING OF MISSING VALUES | |
| 9.3 | HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS 1 | |
| | DATA ANALYSIS | |
| 10.1 | MAIN ANALYSIS 1 | 1 |
| 10.2 | CAPETY ANALYCIC 1 | 7 |
| | SAFETY ANALYSIS | |
| 10. | .3.1 Adverse Events | 0 |
| 11 ( | QUALITY CONTROL2 | |
| | REFERENCES | |
| 12. r | PUBLISHED REFERENCES | |
| 12.1 | FUBLISHED REFERENCES | 4 |

**1199.402** 

#### 1. LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction
ADS Analysis Data Set

ALT Alanine aminotransferase AST Aspartate aminotransferase

BMI Body mass index BSA Body surface area CRF Case Report Form

DMARDs Disease Modifying Anti-Rheumatic Drugs

EDC Electronic Data Capture
FVC Forced Vital Capacity
HLGT High level group term
HLT High level term

HOT Home Oxygen Therapy ILD Interstitial Lung Disease

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed Model Repeated Measures

NIS Non-interventional Study

PD Protocol deviation

PF-ILD Chronic fibrosing Interstitial Lung Diseases with a progressive

phenotype

PMS Post-marketing surveillance

PT Preferred term

RMP Risk Management Plan SMQ Standardised MedDRA query

SOC System organ class TBILI Total bilirubin

SEAP Statistical and Epidemiological Analysis Plan

ULN Upper Limit of Normal

1199.402 

#### 2. RESPONSIBLE PARTIES

Contact details and the list of all investigators will be kept in a stand-alone document. This document will be managed in the Post Marketing Surveillance (PMS) tracking system which manages the contracts with site and investigators name.

#### 3. PURPOSE AND SCOPE

The purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the PMS data.

This SEAP assumes familiarity with the Non-interventional Study (NIS) Protocol, including Protocol Amendments. In particular, the SEAP is based on the planned analysis specification as written in NIS Protocol Section 9.7 "DATA ANALYSIS". Therefore, SEAP readers may consult the NIS Protocol for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size.

#### 4. AMENDMENTS AND UPDATES

| Number | Date | Section of study protocol | Amendment or update | Reason |
|--------|------|---------------------------|---------------------|--------|
| None | | | | |

### 5. RESEARCH QUESTION AND OBJECTIVE

The primary objective is to evaluate the frequency of adverse drug reactions (focus on hepatic function disorders) of Ofev Capsules under the real world setting in patients with PF-ILD.

Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402


#### 6. RESEARCH METHODS

#### 6.1 STUDY DESIGN

This is a non-interventional study based on newly collected data of patients under routine care to confirm safety of Ofev Capsules in the real-world setting in Japanese patients with PF-ILD.

#### 6.2 **SETTING**

#### 6.2.1 **Study sites**

Sites throughout entire country will be equally listed according to the size of the hospitals or general clinics at which Ofev Capsules are available for prescription.

Planned number of sites: Approximately 100 Sites

A medical representative will explain the objective and design of this study to investigators at each study site and conclude a written contract with the head of the study site (e.g., hospital director).

#### Inclusion/ exclusion criteria 6.2.2

#### Inclusion criteria

Patients in Japan with PF-ILD who are prescribed with Ofev Capsules and have never been treated with Ofev Capsules before enrolment will be included.

#### Exclusion criteria

- Diagnosis of IPF
- Patients with PF-ILD due to systemic scleroderma as the underlying disease

#### 6.2.3 Registration period

From October 2020 to September 2022

#### 6.2.4 Patient registration method

The registration method will be a continuous investigation system. Patients who begin treatment with Ofev Capsules after the conclusion of the contract will be registered by entering necessary information in the Electronic Data Capture (EDC) system within 14 days whenever possible from the day of treatment initiation (inclusive).

Patient registration will be stopped when the overall target number of patients for the study is reached. After the end of the registration period, investigators use a signed form to confirm that patients have been registered continuously at the site. A log of all patients included in the study will be maintained at the site.

Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402


#### 6.3 STUDY POPULATION

Provide a table specifying the definition of all important Protocol deviations (PDs) with columns for PD category / code, PD description, additional comment/example and a column to describe which PDs will be used to exclude patients from the different patient analysis sets. The final decision about which patients will be excluded from analysis sets will be taken during the course of the study and at report planning meetings before database lock at the latest.

Table 6.3: 1 Important protocol deviations

| Category /<br>Code | | Description | Requirements | Method | Exclud<br>ed<br>from |
|---|---|---|---|---|---|
| A | | Entrance criteria not met | | | |
| | A1 Patient of non-PF-ILD | | PF-ILD Reason of use is not PF-ILD Automated Patients who correspond the below exclusion criteria | | Effecti<br>veness |
| | | | · Diagnosis of IPF | | |
| | | | Patients with PF-ILD due to<br>systemic scleroderma as the<br>underlying disease | | |
| | A2 | Patient received Ofev ® treatment before registration | See Previous Medication code:3999039 (include 9 digits code) | Automated | Safety/<br>Effecti<br>veness |
| В | | Trial medication | | | |
| | B1 No treatment with Ofev® Capsules | | No treatment status | Automated | Safety/<br>Effecti<br>veness |
| C | | Missing data | | | |
| | C1 | No effectiveness outcomes | No effectiveness outcomes at baseline and/or post treatment (FVC, FVC% predicted, FEV1, FEV1% predicted, DLco% predicted, SpO2 and time to first acute ILD exacerbation) | Automated | Effecti<br>veness |
| D | | Invalid registration | | | |
| | D1 | No patient visit after entry | Administration status is "No visit since the first visit" | Automated | Safety/<br>Effecti<br>veness |
| | D2 Multiple registration D3 Registration rule not followed | | <ul> <li>Pick out patients that falling under all of the following:</li> <li>Sex, birthday, Ofev start date and site name are the same</li> <li>Height is within ± 2 cm</li> <li>Weight is within ± 5 kg</li> </ul> | Manual | Safety/<br>Effecti<br>veness |
| | | | See NIS Protocol section 9.2.2.2 and 9.2.2.3 | Manual | Safety/<br>Effecti<br>veness |
| | | Patient started Ofev ® treatment out of registration period | See NIS Protocol section 9.2.2.2 | Automated | Safety/<br>Effecti<br>veness |

Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402


| ĺ | Cate | egory / | Description | Requirements | Method | Exclud |
|---|---|---|---|---|---|---|
| | Cod | e | | | | ed |
| | | | | | | from |
| ĺ | | D5 | Not continuous investigation | See NIS Protocol section 9.2.2.3 | Manual | Safety/ |
| | | | | | | Effecti |
| | | | | | | veness |

The safety set will be the basis of all demographic, baseline and safety analyses. Effectiveness analysis will be on basis of the effectiveness set.

- Safety set: This patient set includes all patients who didn't have important PDs regarding safety and regulatory issues as marked as "Safety" in Table 6.3: 1.
- Effectiveness set:
  This patient set includes all patients in safety set with PF-ILD and have effectiveness information. (Patients marked "Effectiveness" in <a href="Table 6.3:1">Table 6.3:1</a> should be excluded from effectiveness analysis.)

#### 6.4 STUDY VISITS

The study will consist of a baseline visit and further visits in a 104-week follow-up for patients who have initiated Ofev Capsules treatment.

With regard to effectiveness and safety endpoints, the term "baseline" refers to the last observed measurement before the first administration of Ofev® Capsules. The first date of the administration of Ofev® Capsules is included in "baseline".

Effectiveness analyses will be performed based on calculated visits as shown in <u>Table 6.4: 1</u>. If two or more data points of a patient fall into the same interval, the closest value to the planned day will be selected. If there are two observations which have the same difference in days to the planned day or if there are two observations on the same day, the first value will be used.

Table 6.4: 1 Baseline, time windows and calculated visits

| | | Time window (actual days on treatment) | |
|---|---|---|---|
| Week label | Planned days | Start | End |
| Baseline | 1 | The last observed measurement administration of Ofev® Cap | |
| Week 4 | 28 | 2 | 56 |
| Week 12 | 84 | 57 | 126 |
| Week 24 | 168 | 127 | 210 |
| Week 36 | 252 | 211 | 308 |
| Week 52 | 364 | 309 | 434 |
| Week 72 | 504 | 435 | 546 |
| Week 84 | 588 | 547 | 630 |

# Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402


| | | Time window (actual days on treatment) | |
|---|---|---|---|
| Week label | Planned days | Start | End |
| Week 96 | 672 | 631 | 700 |
| Week 104 | 728 | 701 | End of study |

**1199.402** 

#### 7. VARIABLES

#### 7.1 EXPOSURES

Exposure to Ofev Capsules is estimated as time from the day Ofev Capsules is initiated until the day the drug is last administrated on a patient-level (or the final contact with the patient during the regular observation period).

Patients newly initiating Ofev Capsules will be followed up to 104 weeks.

#### 7.2 OUTCOMES

#### 7.2.1 Primary outcomes

The primary outcome of this study is the frequency of adverse drug reactions (ADRs). There is no primary outcome for effectiveness as the primary objective of a PMS is evaluating safety.

#### 7.2.2 Secondary outcomes

None



#### 7.3 COVARIATES

The covariates included in the model analysis is described in Section 10.2.4.

Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1100 402

**1199.402** 

#### 8. DATA SOURCES

Case Report Forms (CRFs) for individual patients will be provided by the sponsor via the EDC system.

In EDC system, three casebooks will be set:

- Book 1 includes baseline, 4 and 12 weeks.
- Book 2 includes 24, 36 and 52 weeks.
- Book 3 includes 72, 84, 96 and 104 weeks.

The data are to be transmitted immediately after being entered into EDC at 12 weeks (Book 1), 52 weeks (Book 2) and 104 weeks (Book 3) after the start of treatment or at discontinuation.

For any adverse events, the data should be immediately entered into EDC and transmitted.

#### 9. DATA MANAGEMENT AND SOFTWARE/TOOLS

#### 9.1 **SOFTWARE/TOOLS**

SAS<sup>®</sup> Version 9.4 or later will be used for all analyses.

#### 9.2 HANDLING OF MISSING VALUES

Safety:

Missing or incomplete AE dates are imputed according to

Missing or partial date information will be replaced according to following rules.

| YEAR | MONTH | DAY | YMD | DT |
|---|---|---|---|---|
| "Unknown" (tick-box) | | UNKNOWN | | |
| уууу | Null or "Unknown" | Null | Yyyy | yyyy/01/01 |
| уууу | mm | Null or "Unknown" | Yyyymm | yyyy/mm/01 |

#### Effectiveness:

Missing effectiveness data will not be imputed.

Missing or partial date information will be replaced according to safety rules.

Note that in general when tabulating AEs, and/or demographic and baseline characteristics variables reported as unknown will be treated as such; otherwise treated as missing data.

#### 9.3 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS

Outliers will not be excluded from analyses unless otherwise noted.

#### 10. DATA ANALYSIS

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / SD / Min / Q1 / Median / Q3 / Max.

For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles should be preferred to mean, standard deviation, minimum and maximum.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to two decimal places. The category missing will be displayed only if there are actually missing values.

#### 10.1 MAIN ANALYSIS

The analysis of the primary outcomes is described in <u>Section 10.3.1</u>.



Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402




Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402




Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402




Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402




Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402




Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402




#### 10.3 SAFETY ANALYSIS

All safety analyses will be performed on the safety set.

Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402


#### **10.3.1** Adverse Events

Unless otherwise specified, the analyses of adverse events (AEs) will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and NOT on the number of AEs.

Furthermore, for analysis of AE attributes such as duration, severity, etc. multiple AE occurrence data, will be collapsed into AE episodes provided that all of the following applies:

- The same MedDRA lowest level term was reported for the occurrences
- The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence)
- Treatment did not change between the onset of the occurrences OR treatment changed between the onset of the occurrences, but no deterioration was observed for the later occurrence

For further details on summarization of AE data, please refer to

Unless otherwise specified, AE analyses will be performed by AE data from Safety data.

An Adverse Drug reaction (ADR) is defined as an AE for which either the investigator or the sponsor (or both) assess the causal relationship to Ofev® Capsules as "Yes". A serious AE is defined as an AE for which either the investigator or the sponsor (or both) assess the seriousness as "Serious".

The SOCs will be sorted according to the standard sort order specified by European Medicines Agency, PTs will be sorted by frequency (within SOC).

The frequency of patients with the following items will be summarized.

- AEs
- ADRs

• AEs leading to death

Serious AEs

The frequency of patients with the following items will be summarized by primary SOC and PT.

Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402 

| • | AEs |
|---|------|
| • | ADRs |

• AEs leading to death

• Serious AEs




Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402

## $\textbf{BOEHRINGER INGELHEIM Group of Companies} \hspace{0.1cm} \textbf{Global ID:} 228892\_82584\_1.0$

Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402 



Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1199.402



Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1100 402

1199.402 



Statistical and Epidemiological Analysis Plan (SEAP) for BI Trial No: 1100 402

1199.402 

### 11. QUALITY CONTROL

All processes are conducted according to

Appropriate records and documents are stored based on the and these processes are checked by internal self-check.

### 12. REFERENCES

#### 12.1 PUBLISHED REFERENCES

Not applicable.

